CLINICAL TRIAL: NCT07186478
Title: The Potential Development of I-FALMIN as a Phytopharmaca Candidate for Albumin Supplementation Derived From Toman Fish in Patients With Pulmonary Tuberculosis
Brief Title: I-FALMIN Albumin Supplement for Patients With Pulmonary Tuberculosis
Acronym: I-FALMIN TB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Collaborators: RSUP Dr. Wahidin Sudirohusodo (Other)
Responsible Party: Principal Investigator, Prof. dr. Muh. Nasrum Massi, Ph.D., Sp.MK (K), Principal Investigator, Department of Microbiology, Faculty of Medicine, Hasanuddin University, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNHAS-TB-CLINTRIAL-2025; 669/UN4.6.4.5.31./ PP36 / 2024 (Other: Health Research Ethics Committee, Faculty of Medicine, Hasanuddin University); RG.02.05.42.423.01.8.2024.1450 (Other: National Agency of Drug and Food Control of Indonesia (BPOM))
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Tuberculosis; Hypoalbuminemia
Keywords: Pulmonary Tuberculosis; Tuberculosis; Albumin supplement; Hypoalbuminemia; Toman Fish (Channa micropeltes); Phytopharmaceutical; I-FALMIN
MeSH Terms: conditions — Tuberculosis, Pulmonary; Hypoalbuminemia; Tuberculosis | interventions — Drugs, Investigational; Starch

STUDY DESIGN:
Intervention Model Description: Participants with pulmonary tuberculosis will be randomly assigned to two parallel groups. The intervention group will receive standard anti-tuberculosis therapy plus I-FALMIN supplementation, while the control group will receive standard anti-tuberculosis therapy plus a placebo designed to resemble I-FALMIN. Outcomes will be compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and investigators are blinded to group allocation. The placebo is designed to be indistinguishable in appearance, taste, and packaging from the Ifalmin supplement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Investigational Drug (Experimental): Participants will receive the investigational drug according to the study protocol.
  Interventions: Drug: Investigational Drug
- Placebo Comparator: Placebo (Placebo Comparator): Participants will receive placebo identical in appearance to the investigational drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Investigational Drug — IFALMIN® is a standardized herbal preparation derived from Channa micropeltes (ikan toman), containing natural albumin. Administered orally in capsule form at a dose of 500 mg, 2-3 times daily, for 1 day.
  Other Names: IFALMIN (standardized extract from channa micropeltes)
  Arms: Experimental: Investigational Drug
Drug: Placebo — Placebo capsule containing inert ingredients (such as starch/lactose), identical in appearance, size, and color to IFALMIN® capsule. Administered orally in capsule form at a dose of 500 mg, 2-3 times daily, for 1 day.
  Other Names: Starch capsule
  Arms: Placebo Comparator: Placebo

SUMMARY:
This study evaluates the potential of I-FALMIN, a supplement derived from toman fish (Channa micropeltes), as an additional source of albumin in patients with pulmonary tuberculosis. Tuberculosis patients often experience low albumin levels, which may slow down recovery. The purpose of this study is to determine whether giving I-FALMIN as a supplement, in addition to standard tuberculosis treatment, can improve albumin levels and support overall health status. The study will compare outcomes between patients who receive I-FALMIN and those who do not.

DETAILED DESCRIPTION:
ulmonary tuberculosis (TB) remains a major public health problem in Indonesia, with high rates of morbidity and mortality. In addition to lung damage, many TB patients experience low serum albumin levels due to chronic infection, malnutrition, and systemic inflammation. Hypoalbuminemia in TB patients is associated with slower recovery, poorer treatment outcomes, and a higher risk of complications.

I-FALMIN is a natural supplement derived from toman fish (Channa micropeltes), which is rich in albumin and essential amino acids. Previous preclinical and early clinical studies have suggested that albumin extracted from toman fish has potential benefits in improving nutritional status and accelerating recovery in patients with chronic illnesses. However, there is limited evidence on its clinical effectiveness as an adjunctive therapy in pulmonary TB.

This study is designed to evaluate the safety and efficacy of I-FALMIN as a phytopharmaceutical candidate to support nutritional recovery in TB patients. Participants will continue to receive standard anti-tuberculosis therapy according to national guidelines. In addition, the intervention group will receive I-FALMIN supplementation, while the control group will receive standard therapy without the supplement.

The primary objective is to determine whether I-FALMIN supplementation increases serum albumin levels compared to standard care alone. Secondary objectives include assessing improvements in clinical symptoms, body weight, immune response, and overall treatment outcomes. Findings from this study are expected to provide scientific evidence to support the development of I-FALMIN as a phytopharmaceutical product that may benefit TB patients in Indonesia and potentially in other countries with high TB burden.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female participants aged 18-60 years.
* Newly diagnosed tuberculosis (TB) patients based on sputum examination using GeneXpert MTB/RIF with MTB positive (low, moderate, or high) and rifampicin resistance not detected.
* Body Mass Index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m²), categorized according to WHO: <18.5 underweight, 18.5-24.9 normal. Eligible participants are those with BMI below the lower normal threshold (<22.5).
* Will receive standard anti-tuberculosis treatment (OAT) regimen (4FDC) according to body weight.
* Serum albumin level <3.5 g/dL before initiation of treatment.
* Willing to undergo randomization and receive the investigational product for 14 days (3 × 4 tablets daily).
* Willing to undergo scheduled follow-up visits at the hospital (clinical examination, BMI measurement, sputum, and blood sampling) on days 15, 29, 43, and 57, as well as sputum smear examination on day 15 and day 57.
* Willing to comply with the study protocol by signing informed consent.

Exclusion Criteria:

* Confirmed HIV infection.
* Pregnant or breastfeeding women.
* History of drug allergy.
* Comorbid hepatitis.
* Complicated liver cirrhosis.
* Nephrotic syndrome.
* History of hematemesis (vomiting blood).
* Renal failure.
* Burn injury.
* Gastric disorders or intestinal diseases.
* Malignancy (cancer).
* Cardiac disorders.
* History of stroke.
* Allergy to fish protein.
* Pulmonary tuberculosis with extrapulmonary involvement or patients currently hospitalized for TB.
* Prior supplementation with albumin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in serum albumin concentration (g/dL) | Day 0 and Day 15
  Change in serum albumin concentration among participants with baseline albumin < 3.1 g/dL. Serum albumin will be measured at Day 0 and reassessed at Day 15 to determine improvement.
Change in Body Mass Index (kg/m²) | Day 0, Day 15, Day 29, Day 43, and Day 57
  Change in BMI (weight in kg/height in m²) from Day 1 measured at day 15, day 29, day 43, and day 57. Weight was measured with calibrated digital scales and height with a stadiometer. Primary analysis compares the mean change from baseline day 0 to day 57.

SECONDARY OUTCOMES:
Proportion of participants with improved chest X-ray findings | baseline day 0 and End of Study day 57
  Chest X-rays will be evaluated by blinded radiologists. Improvement is defined as reduction in infiltrates or consolidation compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUD Wahidin Sudirohusodo, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data